CLINICAL TRIAL: NCT03475368
Title: Diet, Intestinal Microbiota and Metabolomics: Evaluation of Possible Synergies
Brief Title: Interactions Between Diet, Intestinal Microbiota and Metabolomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gioacchino Leandro, Director of Gastroenterology and Clinical Nutrition, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders | interventions — Diet, Vegetarian; Diet, Mediterranean

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vegetarian diet (Experimental): People randomized to interventional groups will take a vegetarian diet (i.e. without animal products, except milk and eggs)
  Interventions: Other: Vegetarian diet
- Low carbs (Experimental): People randomized to interventional groups will take a low carbs diet (i.e. with a limited amount of carbohydrates).
  Interventions: Other: Low carbs diet
- Mediterranean diet (Active Comparator): People randomized to interventional groups will take a mediterranean diet (i.e. with low glycemic index carbohydrates and vegetables).
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Vegetarian diet — People randomized to this interventional group will take a vegetarian diet (i.e. without animal products, except milk and eggs).
  Arms: Vegetarian diet
Other: Low carbs diet — People randomized to this interventional group will take low carbs diet (i.e. with a limited amount of carbohydrates)
  Arms: Low carbs
Other: Mediterranean diet — People randomized to this interventional group will take a traditional Mediterranean diet.
  Arms: Mediterranean diet

SUMMARY:
It is widely known that the quality of the diet is able to modify the expression of many bacterial genes populating the intestine of the host, as well as the type of bacteria themselves. This is also expressed with a more or less evident and troublesome after meals symptomatology that many patients complain to the health care staff.

A good composition of the microbiota is crucial for the health of the individual, both at the intestinal level as well as at the systemic level because, depending on the type of food substrate available at the intestinal level, metabolites will be produced capable of positively or negatively affect the health of the individual.

In fact, scientific evidence shows the existence of the causal link between the health of the microbiota and the genesis of inflammatory diseases not only intestinal, but also systemic, and even of cancer, obesity, metabolic syndrome and atherosclerosis.

The recent diffusion of gene sequencing techniques has brought significant developments in the study of the human and bacterial genome, which allow to produce enormous quantities of sequences at a lower cost and at a higher speed than previous techniques.

Therefore the clinical Nutrition Clinic of the IRCCS De Bellis in Castellana Grotte (BA) proposes to check if changes in the intestinal microbiota correlate, not only with anthropometric and clinical-laboratory parameters, but also with the typical symptoms of irritable bowel syndrome (IBS), a functional pathology very widespread with the advent of the modern era, in which, a diet rich in sugars and proteins of animal origin and poor in plant foods, is unfortunately common also in the areas of the Mediterranean basin.

ELIGIBILITY:
Inclusion Criteria:

* No major comorbidities with a life expectancy less than 12 months;
* BMI between 29 and 33 kg/m2
* Serum cholesterol 200-260 mg/dl
* Serum triglycerides > 150 mg/dl

Exclusion Criteria:

* Antibiotics or prebiotics in the 3 months before the enrollment;
* Use of statins or other medications for lowering cholesterol;
* Menopause;
* Previous history of cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in weight | At baseline and after two months.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera Specializzata in Gastroenterologia Saverio de Bellis, Castellana Grotte, BARI, Italy

REFERENCES:
- [Background] Zimmer J, Lange B, Frick JS, Sauer H, Zimmermann K, Schwiertz A, Rusch K, Klosterhalfen S, Enck P. A vegan or vegetarian diet substantially alters the human colonic faecal microbiota. Eur J Clin Nutr. 2012 Jan;66(1):53-60. doi: 10.1038/ejcn.2011.141. Epub 2011 Aug 3. PMID 21811294
- [Background] Turnbaugh PJ, Ley RE, Hamady M, Fraser-Liggett CM, Knight R, Gordon JI. The human microbiome project. Nature. 2007 Oct 18;449(7164):804-10. doi: 10.1038/nature06244. PMID 17943116